CLINICAL TRIAL: NCT03316625
Title: Reference Curve on Bone Mineral Density in Young Adult: French Multicenter Study
Acronym: COURDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2016-06
Record Dates: First submitted 2017-09-22; First posted 2017-10-20 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2017-10

CONDITIONS: Bone Mineral Density; Grip Strength; Physical Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone mineral density (Experimental): Bone densitometry measurement : Measurement of bone mineral densitometry with bone densitometry
  Interventions: Diagnostic Test: Bone densitometry measurement

INTERVENTIONS:
Diagnostic Test: Bone densitometry measurement — Bone Densitometry and measurement of body composition

SUMMARY:
In men, the hope of lower life, the absence of equivalent of menopause and the existence of a higher peak bone mass are three factors that explain the lower incidence of osteoporosis in men. Epidemiological data indicate a prevalence of 15% among men aged over 50 years (Szulc et al. 2000). According to global analyzes, the number of fractures of the upper end of the femur in humans will increase from 400 000 to 800 000 per year between 2000 and 2025 (Kanis et al. 2004). Furthermore the mortality due to major osteoporotic fractures when they occur in humans than that seen in women (Johnell and al.2001).The main goal of this study is to establish reference curves in elderly male volunteers from 20 to 30 years through the assessment of bone mineral density of the spine, hip, and the measurement of body composition (fat mass, lean mass). This study will allow us to establish the mean and standard deviation of the value of the young adults of the same sex, which will eventually be applied in the calculation of the "T-score" for older people.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 20 and 30 years
* Caucasians

Exclusion Criteria:

* Lack of informed consent
* Pieces of metal or plastic parts in the field
* Diseases which cause technical difficulties for the correct evaluation of the hip and spine (severe dysplasia, hip surgery or lumbar spine)

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
bone mineral density of the spine | Day 0
  to establish reference curves in elderly male volunteers from 20 to 30 years through the assessment of bone mineral density of the spine, hip, the measurement of body composition (fat mass, lean mass)
bone mineral density of the hip | Day 0
  to establish reference curves in elderly male volunteers from 20 to 30 years through the assessment of bone mineral density of the spine, hip, the measurement of body composition (fat mass, lean mass)
body composition (fat mass, lean mass) | day 0
  to establish reference curves in elderly male volunteers from 20 to 30 years through the assessment of bone mineral density of the spine, hip, the measurement of body composition (fat mass, lean mass)

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSAILLES, Dr, Principal Investigator — CHR Orléans
Locations (3):
- France (3):
  - Chru Lille, Lille
  - CHRU Lyon, Lyon
  - CHR Orléans, Orléans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrahamsen B, Hansen TB, Jensen LB, Hermann AP, Eiken P. Site of osteodensitometry in perimenopausal women: correlation and limits of agreement between anatomic regions. J Bone Miner Res. 1997 Sep;12(9):1471-9. doi: 10.1359/jbmr.1997.12.9.1471. PMID 9286764
- [Background] Ahmed AI, Blake GM, Rymer JM, Fogelman I. Screening for osteopenia and osteoporosis: do the accepted normal ranges lead to overdiagnosis? Osteoporos Int. 1997;7(5):432-8. doi: 10.1007/s001980050029. PMID 9425500
- [Background] Baumgartner RN. Body composition in elderly persons: a critical review of needs and methods. Prog Food Nutr Sci. 1993 Jul-Sep;17(3):223-60. PMID 8234779